CLINICAL TRIAL: NCT02600455
Title: Outline of Use-Results Survey for ORENCIA® Subcutaneous Injection 125mg Syringe 1mL
Brief Title: Use-Results Survey for ORENCIA® Subcutaneous Injection 125mg Syringe 1mL
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-515
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who are treated with ORENCIA: Patients who are treated with ORENCIA according to the approved indications, and dosage and administration
  Interventions: Drug: Orencia

INTERVENTIONS:
Drug: Orencia

SUMMARY:
The purpose of this study to collect information on the safety, especially localized injection site reactions, and efficacy of ORENCIA Subcutaneous Injection 125mg Syringe 1mL in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are beginning to receive the treatment with ORENCIA Subcutaneous Injection 125mg Syringe 1mL under the approved indications, dosage, and administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated with ORENCIA according to the approved indications, and dosage and administration.
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety measured by number of Adverse events and laboratory abnormalities associated with adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx